CLINICAL TRIAL: NCT01592955
Title: Glaucoma Treatment by Cyclo-coagulation Using High Intensity Focused Ultrasound With the EyeOP1 Medical Device.
Brief Title: Glaucoma Treatment by Cyclo-coagulation Using High Intensity Focused Ultrasound (HIFU)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EyeTechCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYEMUST-2
Record Dates: First submitted 2012-05-04; First posted 2012-05-07 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2013-03

CONDITIONS: Glaucoma
Keywords: Glaucoma; Cyclocoagulation; HIFU High Intensity Focused Ultrasound
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EYEOP1 device (Experimental): cyclocoagulation HIFU
  Interventions: Device: EYEOP1

INTERVENTIONS:
Device: EYEOP1 — Cyclocoagulation using High Intensity Focused Ultrasound with EYEOP1 device

SUMMARY:
The purpose of this study is to evaluate the effectiveness and the safety of the cyclocoagulation using High Intensity Focused Ulatrsound with the EYEOP1 device in glaucoma patients

ELIGIBILITY:
Inclusion Criteria:

* Refractory Glaucoma
* IOP > 21 mm Hg
* No previous intraocular surgery or laser treatment during the 90 days before HIFU day
* Age > 18 years
* Informed consent sgned by the subject

Exclusion Criteria:

* Normal Tension Glaucoma
* Glaucoma drainage device implanted and still present in the eye to be treated
* History of ocular or retrobulbar tumor
* Ocular infection within 14 days prior to the HIFU procedure
* Aphakic patient
* Ocular disease other than glaucoma that may affect assessment of visual and/or IOP (choroidal hemorrhage or detachment, lens subluxation, thyroid ophthalmopathy, proliferative diabetic retinopathy, clinical significant macular edema)
* Pregnant or breast-feeding women, or lack of contraception use among women likely to have a child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint : Success / failure rate at 1 year | 12 months
  IOP change (mm Hg and percent) from baseline to 12 months post-HIFU treatment. (Success defined by IOP reduction > 20% compared to the baseline IOP or IOP < 21 mmHg)

SECONDARY OUTCOMES:
Safety measures | 12 months
  Number of device and procedure-related and others complications during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Laurent FARCY, Study Director — EyeTechCare
Locations (7):
- The Sam Rothberg Glaucoma Center, Goldschleger EyeInstitute, Sheba Medical Center, Tel Litwinsky, Israel
- Italy (3):
  - Ospedale San Paolo, Milan
  - Institute Ophthalmology - Universita di Parma, Parma
  - Clinica Oculistica Universitaria - P-O Oftalmico, Torino
- Hospital Clinico San Carlos, Madrid, Spain
- Switzerland (2):
  - Hôpitaux Universitaires de Genève, Geneva
  - Clinique de Montchoisi - Glaucoma center, Lausanne

REFERENCES:
- [Result] Melamed S, Goldenfeld M, Cotlear D, Skaat A, Moroz I. High-intensity focused ultrasound treatment in refractory glaucoma patients: results at 1 year of prospective clinical study. Eur J Ophthalmol. 2015 Nov-Dec;25(6):483-9. doi: 10.5301/ejo.5000620. Epub 2015 May 13. PMID 25982212